CLINICAL TRIAL: NCT04476030
Title: A Phase 3, Randomized, Double-Blind Study Comparing the Efficacy and Safety of SAGE-217 Plus an Antidepressant Versus Placebo Plus an Antidepressant in Adults With Major Depressive Disorder
Brief Title: A Comparative Study of Sage-217 Plus an Antidepressant (ADT) Versus Placebo Plus an ADT in Adults With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 217-MDD-305
Record Dates: First submitted 2020-07-15; First posted 2020-07-17 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Depressive Disorder, Major
Keywords: Major Depressive Disorder; MDD; SAGE-217
MeSH Terms: conditions — Depressive Disorder, Major | interventions — zuranolone; Sertraline; Escitalopram; Citalopram; Duloxetine Hydrochloride; Desvenlafaxine Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo + Assigned ADT (Active Comparator): Participants received SAGE-217-matching placebo capsules, orally, once daily along with an assigned ADT (sertraline, escitalopram, citalopram, duloxetine, or desvenlafaxine administered per labeled prescribing information), daily, from Day 1 through 14, followed by the same ADT, per labeled prescribing information, daily, up to Day 42.
  Interventions: Drug: Matching Placebo; Drug: Sertraline; Drug: Escitalopram; Drug: Citalopram; Drug: Duloxetine; Drug: Desvenlafaxine
- SAGE-217 + Assigned ADT (Experimental): Participants received SAGE-217, 50 milligrams (mg), orally, once daily along with an assigned ADT (sertraline, escitalopram, citalopram, duloxetine, or desvenlafaxine administered per labeled prescribing information), daily from Day 1 through 14, followed by the same ADT, per labeled prescribing information, daily, up to Day 42.
  Interventions: Drug: SAGE-217; Drug: Sertraline; Drug: Escitalopram; Drug: Citalopram; Drug: Duloxetine; Drug: Desvenlafaxine

INTERVENTIONS:
Drug: SAGE-217 — Oral capsules
  Arms: SAGE-217 + Assigned ADT
Drug: Matching Placebo — Oral capsules
  Arms: Placebo + Assigned ADT
Drug: Sertraline — Oral tablets
Drug: Escitalopram — Oral tablets
Drug: Citalopram — Oral tablets
Drug: Duloxetine — Oral capsules
Drug: Desvenlafaxine — Oral tablets

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of SAGE-217 plus an ADT in the treatment of major depressive disorder (MDD) compared to placebo plus an ADT.

DETAILED DESCRIPTION:
This study was previously posted by Sage Therapeutics. In November 2023, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MDD as diagnosed by Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition Clinical Trials Version (SCID-5-CT), with symptoms that have been present for at least a 4-week period
* 17-item Hamilton Rating Scale for Depression (HAM-D-17) total score of ≥24 at Screening and Day 1
* Participant in good physical health and has no clinically significant findings, as determined by the investigator, on physical examination, 12-lead electrocardiogram (ECG), or clinical laboratory tests
* Participant is willing, able, and eligible to take at least 1 of the 5 ADTs specified in the protocol (an eligible ADT is an ADT that has not been taken during the current depressive episode and for which the participant has no contraindications; further, a participant is not eligible for citalopram if escitalopram has been taken during the current depressive episode, and vice versa)

Exclusion Criteria:

* Has attempted suicide associated with the current episode of MDD
* Participant had onset of the current depressive episode during pregnancy or 4 weeks postpartum, or the participant has presented for screening during the 6-month postpartum period
* Participant has treatment-resistant depression
* History of bipolar disorder, schizophrenia, and/or schizoaffective disorder
* Known allergy to SAGE-217, allopregnanolone, or related compounds
* Has taken antidepressants within 30 days prior to Day 1, and/or has taken fluoxetine within 60 days prior to Day 1

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 440 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-12-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (45):
- United States (45):
  - Sage Investigational Site, Dothan, Alabama
  - Sage Investigational Site, Phoenix, Arizona
  - Sage Investigational Site, Anaheim, California
  - Sage Investigational Site, Costa Mesa, California
  - Sage Investigational Site, Glendale, California
  - Sage Investigational Site, Irvine, California
  - Sage Investigational Site, Los Alamitos, California
  - Sage Investigational Site, Oceanside, California
  - Sage Investigational Site, Orange, California
  - Sage Investigational Site, Riverside, California
  - Sage Investigational Site, San Diego, California
  - Sage Investigational Site, Temecula, California
  - Sage Investigational Site, Colorado Springs, Colorado
  - Sage Investigational Site, Cromwell, Connecticut
  - Sage Investigational Site, Norwich, Connecticut
  - Sage Investigational Site, Coral Springs, Florida
  - Sage Investigational Site, Jacksonville, Florida
  - Sage Investigational Site, Orlando, Florida
  - Sage Investigational Site, Pensacola, Florida
  - Sage Investigational Site, Alpharetta, Georgia
  - Sage Investigational Site, Atlanta, Georgia
  - Sage Investigational Site, Marietta, Georgia
  - Sage Investigational Site, Savannah, Georgia
  - Sage Investigational Site, Chicago, Illinois
  - Sage Investigational Site, Towson, Maryland
  - Sage Investigational Site, Watertown, Massachusetts
  - Sage Investigational Site, Ann Arbor, Michigan
  - Sage Investigational Site, Saint Charles, Missouri
  - Sage Investigational Site, Lincoln, Nebraska
  - Sage Investigational Site, Cherry Hill, New Jersey
  - Sage Investigational Site, Marlton, New Jersey
  - Sage Investigational Site, Princeton, New Jersey
  - Sage Investigational Site, Albuquerque, New Mexico
  - Sage Investigational Site, Brooklyn, New York
  - Sage Investigational Site, Mount Kisco, New York
  - Sage Investigational Site, Beachwood, Ohio
  - Sage Investigational Site, Cincinnati, Ohio
  - Sage Investigational Site, North Canton, Ohio
  - Sage Investigational Site, Oklahoma City, Oklahoma
  - Sage Investigational Site, Plymouth Meeting, Pennsylvania
  - Sage Investigational Site, Austin, Texas
  - Sage Investigational Site, Dallas, Texas
  - Sage Investigational Site, Houston, Texas
  - Sage Investigational Site, Wichita Falls, Texas
  - Sage Investigational Site, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Parikh SV, Aaronson ST, Mathew SJ, Alva G, DeBattista C, Kanes S, Lasser R, Bullock A, Kotecha M, Jung J, Forrestal F, Jonas J, Vera T, Leclair B, Doherty J. Efficacy and safety of zuranolone co-initiated with an antidepressant in adults with major depressive disorder: results from the phase 3 CORAL study. Neuropsychopharmacology. 2024 Jan;49(2):467-475. doi: 10.1038/s41386-023-01751-9. Epub 2023 Oct 24. PMID 37875578

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 53 investigative sites in the United States from 9 November 2020 to 22 December 2021.
Pre-assignment Details: A total of 440 participants were enrolled in the study of which 430 participants received at least 1 dose of the assigned treatment. The study consisted of a 28-day Screening period, a 14-day Double-blind Treatment Period, and a 28-day antidepressant therapy (ADT) continuation period.
Period: Overall Study
Arm/Group | Placebo + Assigned ADT | SAGE-217 + Assigned ADT
Started | 220 | 220
Safety Population (Safety Set included all participants who administered blinded IP.) | 218 | 212
Completed | 177 | 180
Not Completed | 43 | 40
Not completed — Withdrawal by Subject | 20 | 16
Not completed — Adverse Event | 10 | 11
Not completed — Lost to Follow-up | 7 | 4
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Deviation | 2 | 0
Not completed — Non-compliance with Investigational Product (IP) | 1 | 0
Not completed — Randomized but not Dosed | 2 | 8

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who administered blinded IP.
Groups:
- SAGE-217 + Assigned ADT: Participants received SAGE-217, 50 mg, orally, once daily along with an assigned ADT (sertraline, escitalopram, citalopram, duloxetine, or desvenlafaxine administered per labeled prescribing information), daily from Day 1 through 14, followed by the same ADT, per labeled prescribing information, daily, up to Day 42.
- Total: Total of all reporting groups
Arm/Group | Placebo + Assigned ADT | SAGE-217 + Assigned ADT | Total
Number analyzed (Participants) | 218 | 212 | 430
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (12.28) | 38.6 (12.72) | 38.1 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 129 | 269
  Male | 78 | 83 | 161
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52 | 41 | 93
  Not Hispanic or Latino | 166 | 171 | 337
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 168 | 153 | 321
  Black or African-American | 31 | 46 | 77
  Asian | 12 | 6 | 18
  Other | 3 | 3 | 6
  More than one race | 4 | 2 | 6
  American-Indian or Alaska Native | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
17-item Hamilton Rating Scale for Depression (HAMD-17) Total Score [Mean (Standard Deviation); unit: score on a scale] — The 17-item HAM-D scale is used to assess the severity of depression. It is comprised of individual ratings related to following symptoms: depressed mood, feelings of guilt, suicide, insomnia, work and activities, retardation, agitation, anxiety, somatic symptoms, genital symptoms, hypochondriasis, loss of weight, and insight. Individual items are scored on either 3-point (0=none to 2=severe) or 5-point scale (0=none/absent to 4=most severe). Total score is the sum of individual items, ranging from 0 (not depressed) to 52 (severely depressed); where a higher score indicates more depression.
  score on a scale | 26.6 (2.58) | 26.8 (2.51) | 26.7 (2.54)
Clinical Global Impression - Severity (CGI-S) Score [Mean (Standard Deviation); unit: score on a scale] — The CGI-S uses a 7-point Likert scale to rate the severity of the participant's illness at the time of assessment, relative to the clinician's past experience with participants who have the same diagnosis. Considering total clinical experience, the investigator rated the participant on severity of mental illness at the time of rating as: 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = extremely ill. A higher score indicated extreme illness.
  score on a scale | 4.9 (0.57) | 5.0 (0.54) | 4.9 (0.55)
Hamilton Anxiety Rating Scale (HAM-A) Total Score [Mean (Standard Deviation); unit: score on a scale] — Each of the 14 items in the HAM-A was defined by a series of symptoms, and measured both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints). The HAM-A total score was calculated as sum of the 14 individual item scores, each rated on a five point scale ranging from 0 (not present) to 4 (very severe). The total score (sum of all individual items) range from 0 to 56, where <17 indicated mild severity, 18 to 24 indicated mild to moderate severity, and 25 to 30 indicated moderate to severe severity. Higher scores indicated more severe disease.
  score on a scale | 20.4 (5.80) | 19.9 (5.28) | 20.1 (5.55)
Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score [Mean (Standard Deviation); unit: score on a scale] — The MADRS is a 10-item diagnostic questionnaire used to measure the severity of depressive episodes in participants with mood disorders. The MADRS total score was calculated as the sum of the 10 individual item scores. Each item yields a score of 0 (no symptoms) to 6 (symptoms of maximum severity). The total MADRS score (sum of all individual items) ranges from 0 (symptoms absent) to 60 (severe depression). Higher MADRS scores indicated more severe depression.
  score on a scale | 34.9 (4.89) | 35.2 (4.70) | 35.0 (4.80)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the HAMD-17 Total Score at Day 3
Description: The 17-item HAM-D scale is used to assess the severity of depression. It is comprised of individual ratings related to following symptoms: depressed mood, feelings of guilt, suicide, insomnia, work and activities, retardation, agitation, anxiety, somatic symptoms, genital symptoms, hypochondriasis, loss of weight, and insight. Individual items are scored on either 3-point (0=none to 2=severe) or 5-point scale (0=none/absent to 4=most severe). Total score is the sum of individual items, ranging from 0 (not depressed) to 52 (severely depressed); where a higher score indicates more depression. A negative change from baseline indicated improvement. Least Squares (LS) mean was estimated using mixed effects model for repeated measures (MMRM) analysis.
Time Frame: Baseline, Day 3
Population: Full analysis set included all randomized participants who administered blinded IP with a valid baseline total score and at least 1 valid postbaseline total score in at least 1 of HAMD-17, HAM-A, MADRS, 9-item Patient Health Questionnaire (PHQ-9) or had a valid baseline and at least 1 valid postbaseline value in at least 1 of CGI-S or Clinical Global Impression - Improvement (CGI-I) score. Overall number of participants analyzed is the number of participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + Assigned ADT | SAGE-217 + Assigned ADT
Number analyzed (Participants) | 210 | 204
score on a scale | -7.0 (0.38) | -8.9 (0.39)
Statistical Analysis 1: Comparison: Placebo + Assigned ADT vs SAGE-217 + Assigned ADT; Test type: Superiority; p = 0.0004, MMRM; LS Mean Difference = -1.9, 95% CI 2-sided [-3.0 to -0.9], Standard Error of Mean 0.55 — Model used was the MMRM with treatment, baseline HAMD-17 total score, antidepressant use (SSRI/SNRI), assessment time point, and time point-by-treatment interaction as fixed effects with unstructured covariance structure

2. Secondary Outcome: Change From Baseline in the HAMD-17 Total Score Over the Double-Blind Treatment Period
Description: The 17-item HAM-D scale is used to assess the severity of depression. It is comprised of individual ratings related to following symptoms: depressed mood, feelings of guilt, suicide, insomnia, work and activities, retardation, agitation, anxiety, somatic symptoms, genital symptoms, hypochondriasis, loss of weight, and insight. Individual items are scored on either 3-point (0=none to 2=severe) or 5-point scale (0=none/absent to 4=most severe). Total score is the sum of individual items, ranging from 0 (not depressed) to 52 (severely depressed); where a higher score indicates more depression. A negative change from baseline indicated improvement. LS mean was estimated using MMRM analysis. The data reported is summary of data collected and analyzed during double-blind treatment period at Baseline, Day 3, Day 8, Day 12, and Day 15 using equal weights for the scheduled visits.
Time Frame: Baseline through Day 15
Population: Full analysis set included all randomized participants who administered blinded IP with a valid baseline total score and at least 1 valid postbaseline total score in at least 1 of HAMD-17, HAM-A, MADRS, PHQ-9 or had a valid baseline and at least 1 valid postbaseline value in at least 1 of CGI-S or CGI-I score.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + Assigned ADT | SAGE-217 + Assigned ADT
Number analyzed (Participants) | 215 | 210
score on a scale | -10.1 (0.39) | -11.7 (0.40)
Statistical Analysis 1: Comparison: Placebo + Assigned ADT vs SAGE-217 + Assigned ADT; Test type: Superiority; p = 0.0054, MMRM; LS Mean Difference = -1.6, 95% CI 2-sided [-2.7 to -0.5], Standard Error of Mean 0.56 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in the HAMD-17 Total Score at Days 15 and 42
Description: The 17-item HAM-D scale is used to assess the severity of depression. It is comprised of individual ratings related to following symptoms: depressed mood, feelings of guilt, suicide, insomnia, work and activities, retardation, agitation, anxiety, somatic symptoms, genital symptoms, hypochondriasis, loss of weight, and insight. Individual items are scored on either 3-point (0=none to 2=severe) or 5-point scale (0=none/absent to 4=most severe). Total score is the sum of individual items, ranging from 0 (not depressed) to 52 (severely depressed); where a higher score indicates more depression. A negative change from baseline indicated improvement. LS mean was estimated using MMRM analysis. The missing values were imputed for the analysis.
Time Frame: Baseline, Days 15 and 42
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + Assigned ADT | SAGE-217 + Assigned ADT
Number analyzed (Participants) | 215 | 210
score on a scale
  Day 15 | -12.9 (0.49) | -13.7 (0.50)
  Day 42 | -14.9 (0.56) | -14.9 (0.56)
Statistical Analysis 1: Comparison: Placebo + Assigned ADT vs SAGE-217 + Assigned ADT; Day 15; Test type: Superiority; p = 0.2477, MMRM; LS Mean Difference = -0.8, 95% CI 2-sided [-2.2 to 0.6], Standard Error of Mean 0.70 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo + Assigned ADT vs SAGE-217 + Assigned ADT; Day 42; Test type: Superiority; p = 0.9248, MMRM; LS Mean Difference = -0.1, 95% CI 2-sided [-1.6 to 1.5], Standard Error of Mean 0.79 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in the HAMD-17 Total Score Around End of Blinded Treatment
Description: The 17-item HAM-D scale is used to assess the severity of depression. It is comprised of individual ratings related to following symptoms: depressed mood, feelings of guilt, suicide, insomnia, work and activities, retardation, agitation, anxiety, somatic symptoms, genital symptoms, hypochondriasis, loss of weight, and insight. Individual items are scored on either 3-point (0=none to 2=severe) or 5-point scale (0=none/absent to 4=most severe). Total score is the sum of individual items, ranging from 0 (not depressed) to 52 (severely depressed); where a higher score indicates more depression. A negative change from baseline indicated improvement. End of blinded treatment was defined as the average of change from baseline values of Days 12, 15 and 18. LS mean was estimated using MMRM analysis.
Time Frame: Baseline, End of blinded treatment assessment (i.e., average of Days 12, 15 , and 18)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + Assigned ADT | SAGE-217 + Assigned ADT
Number analyzed (Participants) | 215 | 210
score on a scale | -12.7 (0.45) | -13.2 (0.46)
Statistical Analysis 1: Comparison: Placebo + Assigned ADT vs SAGE-217 + Assigned ADT; Test type: Superiority; p = 0.4458, MMRM; LS Mean Difference = -0.5, 95% CI 2-sided [-1.8 to 0.8], Standard Error of Mean 0.65 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Participants With HAMD-17 Response at Day 15 and Day 42
Description: HAM-D response was defined as having a 50% or greater reduction from baseline in HAM-D total score. The 17-item HAM-D scale is used to assess the severity of depression. It is comprised of individual ratings related to following symptoms: depressed mood, feelings of guilt, suicide, insomnia, work and activities, retardation, agitation, anxiety, somatic symptoms, genital symptoms, hypochondriasis, loss of weight, and insight. Individual items are scored on either 3-point (0=none to 2=severe) or 5-point scale (0=none/absent to 4=most severe). Total score is the sum of individual items, ranging from 0 (not depressed) to 52 (severely depressed); where a higher score indicates more depression. Percentages were rounded off to the first decimal point.
Time Frame: At Days 15 and 42
Population: Full analysis set included all randomized participants who administered blinded IP with a valid baseline total score and at least 1 valid postbaseline total score in at least 1 of HAMD-17, HAM-A, MADRS, PHQ-9 or had a valid baseline and at least 1 valid postbaseline value in at least 1 of CGI-S or CGI-I score. Number analyzed is the number of participants with data available for analysis at the specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Assigned ADT | SAGE-217 + Assigned ADT
Number analyzed (Participants) | 215 | 210
percentage of participants
  Day 15: number analyzed (Participants) | 197 | 189
  Day 15 | 49.2 | 53.4
  Day 42: number analyzed (Participants) | 176 | 177
  Day 42 | 65.3 | 59.9
Statistical Analysis 1: Comparison: Placebo + Assigned ADT vs SAGE-217 + Assigned ADT; Day 15; Test type: Superiority; p = 0.4946, Binary Response Model; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.78 to 1.69] — GEE for binary response model was used with factors for treatment, baseline HAMD-17 total score, antidepressant use (SSRI/SNRI), assessment time point, and time point-by-treatment interaction with unstructured covariance structure; Generalized estimating equation is abbreviated as GEE in the method of estimation section
Statistical Analysis 2: Comparison: Placebo + Assigned ADT vs SAGE-217 + Assigned ADT; Day 42; Test type: Superiority; p = 0.3579, Binary Response Model; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.55 to 1.24] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Percentage of Participants With HAMD-17 Remission at Day 15 and Day 42
Description: HAM-D remission was defined as having a HAM-D total score of ≤7. The 17-item HAM-D scale is used to assess the severity of depression. It is comprised of individual ratings related to following symptoms: depressed mood, feelings of guilt, suicide, insomnia, work and activities, retardation, agitation, anxiety, somatic symptoms, genital symptoms, hypochondriasis, loss of weight, and insight. Individual items are scored on either 3-point (0=none to 2=severe) or 5-point scale (0=none/absent to 4=most severe). Total score is the sum of individual items, ranging from 0 (not depressed) to 52 (severely depressed); where a higher score indicates more depression. Percentages were rounded off to the first decimal point.
Time Frame: Days 15 and 42
Population: Full analysis set included all randomized participants who administered blinded IP with a valid baseline total score and at least 1 valid postbaseline total score in at least 1 of HAMD-17, HAM-A, MADRS, PHQ-9 or had a valid baseline and at least 1 valid postbaseline value in at least 1 of CGI-S or CGI-I score. Number analyzed is number of participants with data available for analysis at the specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Assigned ADT | SAGE-217 + Assigned ADT
Number analyzed (Participants) | 215 | 210
percentage of participants
  Day 15: number analyzed (Participants) | 197 | 189
  Day 15 | 21.8 | 29.1
  Day 42: number analyzed (Participants) | 176 | 177
  Day 42 | 39.2 | 37.9
Statistical Analysis 1: Comparison: Placebo + Assigned ADT vs SAGE-217 + Assigned ADT; Day 15; Test type: Superiority; p = 0.1417, Binary Response Model; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.89 to 2.24] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Placebo + Assigned ADT vs SAGE-217 + Assigned ADT; Day 42; Test type: Superiority; p = 0.7872, Binary Response Model; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.62 to 1.44] — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Change From Baseline in CGI-S Score at Day 15
Description: The CGI-S uses a 7-point Likert scale to rate the severity of the participant's illness at the time of assessment, relative to the clinician's past experience with participants who have the same diagnosis. Considering total clinical experience, the investigator rated the participant on severity of mental illness at the time of rating as: 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = extremely ill. A higher score indicated extreme illness. A negative change from baseline indicated improvement. LS mean was estimated using MMRM analysis.
Time Frame: Baseline and Day 15
Population: Full analysis set included all randomized participants who administered blinded IP with a valid baseline total score and at least 1 valid postbaseline total score in at least 1 of HAMD-17, HAM-A, MADRS, PHQ-9 or had a valid baseline and at least 1 valid postbaseline value in at least 1 of CGI-S or CGI-I score. Overall number of participants analyzed is the number of participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Active Comparator: Placebo + Assigned ADT: Participants received SAGE-217-matching placebo capsules, orally, once daily along with an assigned ADT (sertraline, escitalopram, citalopram, duloxetine, or desvenlafaxine administered per labeled prescribing information), daily, from Day 1 through 14, followed by the same ADT, per labeled prescribing information, daily, up to Day 42.
- Experimental: SAGE-217 + Assigned ADT: Participants received SAGE-217, 50 mg, orally, once daily along with an assigned ADT (sertraline, escitalopram, citalopram, duloxetine, or desvenlafaxine administered per labeled prescribing information), daily from Day 1 through 14, followed by the same ADT, per labeled prescribing information, daily, up to Day 42.
Arm/Group | Active Comparator: Placebo + Assigned ADT | Experimental: SAGE-217 + Assigned ADT
Number analyzed (Participants) | 197 | 189
score on a scale | -1.7 (0.09) | -1.9 (0.09)
Statistical Analysis 1: Comparison: Active Comparator: Placebo + Assigned ADT vs Experimental: SAGE-217 + Assigned ADT; Test type: Superiority; p = 0.1993, MMRM; LS Mean Difference = -0.2, 95% CI 2-sided [-0.4 to 0.1], Standard Error of Mean 0.13 — Model used was the MMRM with treatment, baseline CGI-S score, antidepressant use (SSRI/SNRI), assessment time point, and time point-by-treatment interaction as fixed effects with unstructured covariance structure

8. Secondary Outcome: Percentage of Participants With CGI-I Response, at Day 3 and Day 15
Description: CGI-I response was defined as having a CGI-I score of "very much improved" or "much improved." The CGI-I employs a 7-point Likert scale to measure the overall improvement in the participant's condition post-treatment. The investigator rated the participant's total improvement whether or not it was due entirely to IP. Response choices included: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. By definition, all CGI-I assessments are evaluated against baseline conditions. Higher scores indicated worse condition. Percentages were rounded off to the first decimal point.
Time Frame: Days 3 and 15
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Assigned ADT | SAGE-217 + Assigned ADT
Number analyzed (Participants) | 215 | 210
percentage of participants
  Day 3: number analyzed (Participants) | 210 | 205
  Day 3 | 12.9 | 22.9
  Day 15: number analyzed (Participants) | 197 | 189
  Day 15 | 54.3 | 56.6
Statistical Analysis 1: Comparison: Placebo + Assigned ADT vs SAGE-217 + Assigned ADT; Day 3; Test type: Superiority; p = 0.0079, Binary Response Model; Odds Ratio (OR) = 2.05, 95% CI 2-sided [1.21 to 3.47] — GEE for binary response model was used with factors for treatment, baseline CGI-S score, antidepressant use (SSRI/SNRI), assessment time point, and time point-by-treatment interaction with unstructured covariance structure
Statistical Analysis 2: Comparison: Placebo + Assigned ADT vs SAGE-217 + Assigned ADT; Day 15; Test type: Superiority; p = 0.6588, Binary Response Model; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.74 to 1.62] — [estimate comment as in outcome 8, analysis 1]

9. Secondary Outcome: Change From Baseline in MADRS Total Score at Day 15
Description: The MADRS is a 10-item diagnostic questionnaire used to measure the severity of depressive episodes in participants with mood disorders. The MADRS total score was calculated as the sum of the 10 individual item scores. Each item yields a score of 0 (no symptoms) to 6 (symptoms of maximum severity). The total MADRS score (sum of all individual items) ranges from 0 (symptoms absent) to 60 (severe depression). Higher MADRS scores indicated more severe depression. A negative change from baseline indicated improvement. LS mean was estimated using MMRM analysis.
Time Frame: Baseline and Day 15
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + Assigned ADT | SAGE-217 + Assigned ADT
Number analyzed (Participants) | 197 | 188
score on a scale | -15.9 (0.75) | -17.2 (0.76)
Statistical Analysis 1: Comparison: Placebo + Assigned ADT vs SAGE-217 + Assigned ADT; Test type: Superiority; p = 0.2322, MMRM; LS Mean Difference = -1.3, 95% CI 2-sided [-3.4 to 0.8], Standard Error of Mean 1.06 — Model used was the MMRM with treatment, baseline MADRS total score, antidepressant use (SSRI/SNRI), assessment time point, and time point-by-treatment interaction as fixed effects with unstructured covariance structure

10. Secondary Outcome: Percentage of Participants With MADRS Response at Day 15
Description: MADRS response was defined as having a 50% or greater reduction from baseline in MADRS total score. The MADRS is a 10-item diagnostic questionnaire used to measure the severity of depressive episodes in participants with mood disorders. The MADRS total score was calculated as the sum of the 10 individual item scores. Each item yields a score of 0 (no symptoms) to 6 (symptoms of maximum severity). The total MADRS score (sum of all individual items) ranges from 0 (symptoms absent) to 60 (severe depression). Higher MADRS scores indicated more severe depression. Percentages were rounded off to the first decimal point.
Time Frame: Day 15
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Assigned ADT | SAGE-217 + Assigned ADT
Number analyzed (Participants) | 197 | 188
percentage of participants | 48.2 | 51.6
Statistical Analysis 1: Comparison: Placebo + Assigned ADT vs SAGE-217 + Assigned ADT; Test type: Superiority; p = 0.5439, Binary Response Model; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.76 to 1.68] — GEE for binary response model was used with factors for treatment, baseline MADRS total score, antidepressant use (SSRI/SNRI), assessment time point, and time point-by-treatment interaction with unstructured covariance structure

11. Secondary Outcome: Percentage of Participants With MADRS Remission at Day 15
Description: MADRS remission was defined as having a MADRS total score of ≤10. The MADRS is a 10-item diagnostic questionnaire used to measure the severity of depressive episodes in participants with mood disorders. The MADRS total score was calculated as the sum of the 10 individual item scores. Each item yields a score of 0 (no symptoms) to 6 (symptoms of maximum severity). The total MADRS score (sum of all individual items) ranges from 0 (symptoms absent) to 60 (severe depression). Higher MADRS scores indicated more severe depression. Percentages were rounded off to the first decimal point.
Time Frame: Day 15
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Assigned ADT | SAGE-217 + Assigned ADT
Number analyzed (Participants) | 197 | 188
percentage of participants | 28.4 | 30.9
Statistical Analysis 1: Comparison: Placebo + Assigned ADT vs SAGE-217 + Assigned ADT; Test type: Superiority; p = 0.7054, Binary Response Model; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.70 to 1.69] — [estimate comment as in outcome 10, analysis 1]

12. Secondary Outcome: Change From Baseline in HAM-A Total Score at Day 15
Description: Each of the 14 items in the HAM-A was defined by a series of symptoms, and measured both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints). The HAM-A total score was calculated as sum of the 14 individual item scores, each rated on a five point scale ranging from 0 (not present) to 4 (very severe). The total score (sum of all individual items) range from 0 to 56, where <17 indicated mild severity, 18 to 24 indicated mild to moderate severity, and 25 to 30 indicated moderate to severe severity. Higher scores indicated more severe disease. Negative change from baseline indicated improvement. LS mean was estimated using MMRM analysis.
Time Frame: Baseline, Day 15
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + Assigned ADT | SAGE-217 + Assigned ADT
Number analyzed (Participants) | 197 | 188
score on a scale | -9.0 (0.44) | -9.5 (0.44)
Statistical Analysis 1: Comparison: Placebo + Assigned ADT vs SAGE-217 + Assigned ADT; Test type: Superiority; p = 0.4188, MMRM; LS Mean Difference = -0.5, 95% CI 2-sided [-1.7 to 0.7], Standard Error of Mean 0.62 — Model used was the MMRM with treatment, baseline HAM-A total score, antidepressant use (SSRI/SNRI), assessment time point, and time point-by-treatment interaction as fixed effects with unstructured covariance structure

13. Secondary Outcome: Time to First HAMD-17 Response
Description: HAM-D response was defined as having a 50% or greater reduction from baseline in HAM-D total score. The 17-item HAM-D scale is used to assess the severity of depression. It is comprised of individual ratings related to following symptoms: depressed mood, feelings of guilt, suicide, insomnia, work and activities, retardation, agitation, anxiety, somatic symptoms, genital symptoms, hypochondriasis, loss of weight, and insight. Individual items are scored on either 3-point (0=none to 2=severe) or 5-point scale (0=none/absent to 4=most severe). Total score is the sum of individual items, ranging from 0 (not depressed) to 52 (severely depressed); where a higher score indicates more depression. Time (in days) from first dose of study drug to time of first HAMD response was reported in this outcome measure.
Time Frame: From first dose of study drug up to first HAMD-17 response (up to approximately 65 days)
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | Placebo + Assigned ADT | SAGE-217 + Assigned ADT
Number analyzed (Participants) | 215 | 210
days | 15 [2 to 50] | 13 [2 to 61]

14. Secondary Outcome: Change From Baseline in Depressive Symptoms at Day 15, as Assessed by PHQ-9
Description: The PHQ-9 is a participant-rated depressive symptom severity scale. The PHQ-9 total score is calculated as the sum of the 9 individual item scores. For individual items, scoring is based on responses to specific questions, as follows: 0 = not at all; 1 = several days; 2 = more than half the days; and 3 = nearly every day. The PHQ-9 possible total score range is 0 to 27, with higher scores reflecting greater depressive symptoms, and is categorized as follows: 0 to 4 = minimal depression, 5 to 9 = mild depression, 10 to 14 = moderate depression, 15 to 19 = moderately severe depression, and 20 to 27 = severe depression. Negative change from baseline indicated improvement. LS mean was estimated using MMRM analysis.
Time Frame: Baseline and Day 15
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + Assigned ADT | SAGE-217 + Assigned ADT
Number analyzed (Participants) | 196 | 188
score on a scale | -8.7 (0.44) | -8.9 (0.44)
Statistical Analysis 1: Comparison: Placebo + Assigned ADT vs SAGE-217 + Assigned ADT; Test type: Superiority; p = 0.7758, MMRM; LS Mean Difference = -0.2, 95% CI 2-sided [-1.4 to 1.0], Standard Error of Mean 0.62 — Model used was the MMRM with treatment, baseline PHQ-9 total score, antidepressant use (SSRI/SNRI), assessment time point, and time point-by-treatment interaction as fixed effects with unstructured covariance structure

15. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal (investigational) product whether or not related to the medicinal (investigational) product. A TEAE was defined as an AE with onset after the start of IP, or any worsening of a pre-existing medical condition/AE with onset after the start of IP and throughout the study.
Time Frame: Up to approximately 58 weeks
Population: Safety Set was defined as all participants who administered blinded IP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Assigned ADT | SAGE-217 + Assigned ADT
Number analyzed (Participants) | 218 | 212
percentage of participants | 65.6 | 74.1

16. Secondary Outcome: Percentage of Participants With TEAEs, Graded by Severity
Description: An AE was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal (investigational) product whether or not related to the medicinal (investigational) product. A TEAE was defined as an AE with onset after the start of IP, or any worsening of a pre-existing medical condition/AE with onset after the start of IP and throughout the study. The severity was graded as mild, moderate and severe.
Time Frame: Up to approximately 58 weeks
Population: Safety Set was defined as all participants who administered blinded IP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Assigned ADT | SAGE-217 + Assigned ADT
Number analyzed (Participants) | 218 | 212
percentage of participants
  Mild | 38.1 | 35.8
  Moderate | 25.2 | 34.4
  Severe | 2.3 | 3.8

ADVERSE EVENTS:
Time Frame: Up to approximately 58 weeks
Description: The All-cause mortality is reported for all randomized participants and serious and other adverse events are reported for safety set that included all participants who administered blinded IP.
Groups:
- Placebo + Assigned ADT: Participants received SAGE-217-matching placebo capsules, orally, once daily aong with an assigned ADT (sertraline, escitalopram, citalopram, duloxetine, or desvenlafaxine administered per labeled prescribing information), daily, from Day 1 through 14, followed by the same ADT, per labeled prescribing information, daily, up to Day 42.
Arm/Group | Placebo + Assigned ADT | SAGE-217 + Assigned ADT
All-Cause Mortality (participants affected / at risk) | 0/220 | 0/220
Serious Adverse Events (participants affected / at risk) | 0/218 | 2/212
Other Adverse Events (participants affected / at risk) | 113/218 | 123/212
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Assigned ADT (N=218) | SAGE-217 + Assigned ADT (N=212)
Seizure like phenomena (Nervous system disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Assigned ADT (N=218) | SAGE-217 + Assigned ADT (N=212)
Somnolence (Nervous system disorders) | 18 | 39
Dizziness (Nervous system disorders) | 16 | 28
Headache (Nervous system disorders) | 32 | 25
Sedation (Nervous system disorders) | 6 | 12
Tremor (Nervous system disorders) | 3 | 11
Dry mouth (Gastrointestinal disorders) | 19 | 20
Nausea (Gastrointestinal disorders) | 51 | 19
Diarrhoea (Gastrointestinal disorders) | 21 | 13
Insomnia (Psychiatric disorders) | 17 | 21
Fatigue (General disorders) | 11 | 18
Decreased appetite (Metabolism and nutrition disorders) | 7 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for non-commercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT04476030/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/30/NCT04476030/SAP_001.pdf